CLINICAL TRIAL: NCT05384171
Title: Measurement-Based Transition Assistance (MBTA): Evaluating the Promise of a Web-Based Approach to Promote Veterans' Support Seeking
Brief Title: Develop and Validation of Measurement-Based Transition Assistance
Acronym: MBTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SDR 21-075
Record Dates: First submitted 2022-03-18; First posted 2022-05-20 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Well-being
Keywords: well-being; mental health; help-seeking; veteran
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants are randomized to an assessment only condition or to the full MBTA intervention (assessment, feedback and resource recommendations)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): MBTA, MBTA satisfaction measures, and other assessment measures at T1 (baseline); MBTA and other assessment measures at T2 (three month follow-up)
  Interventions: Behavioral: Measurement-Based Transition Assistance (MBTA)
- Active Control Group (Active Comparator): assessment measures only at T1 (baseline); MBTA, MBTA satisfaction measures, and other assessment measures at T2 (three month follow-up)
  Interventions: Behavioral: Measurement-Based Transition Assistance (MBTA)

INTERVENTIONS:
Behavioral: Measurement-Based Transition Assistance (MBTA) — Measurement-Based Transition Assistance (MBTA) asks Veterans about their well-being and then provides Veterans with individualized feedback on areas in which they would benefit from additional support with regard to their health, vocational, financial, and social circumstances, along with personalized recommendations for relevant programs, services, and supports.

SUMMARY:
Although some Veterans seek help when they experience post-military readjustment challenges, many do not. One factor that stands in the way of Veterans' willingness to seek help for these challenges is their lack of knowledge, both with regard to how severe challenges must be to warrant help-seeking and what resources are available to address these challenges. Measurement-Based Transition Assistance (MBTA) aims to address these barriers to help-seeking by providing Veterans with individualized feedback on areas in which they would benefit from additional support with regard to their health, vocational, financial, and social circumstances, along with personalized recommendations for relevant programs, services, and supports. If effective, this scalable, population-based intervention strategy could be used independently or in conjunction with other approaches to enhancing Veterans' help-seeking to interrupt high-risk trajectories before they lead to chronic maladjustment and increased risk for suicide.

DETAILED DESCRIPTION:
Background: There is a growing recognition that Veterans' broader vocational, financial, and social circumstances have substantial implications for their health and health care. These circumstances include factors such as whether a Veteran has a job, can pay his or her bills, and has a strong social support network. Although some Veterans seek help when they experience challenges in these life domains, many do not. One factor that stands in the way of Veterans' help-seeking is lack of knowledge, both with regard to how severe challenges must be to warrant help-seeking and what resources are available to address these challenges. If not addressed, Veterans' readjustment challenges may become chronic, escalate in severity, and negatively influence more aspects of Veterans' lives over time and thus, become more difficult to intervene on.

Significance: This study will provide a preliminary examination of the potential benefit of Measurement-Based Transition Assistance (MBTA) in promoting Veterans' help-seeking. MBTA involves providing individualized feedback on areas in which Veterans would benefit from additional support, along with personalized recommendations for relevant programs, services, and supports. If effective, this scalable, population-based intervention strategy could be used independently or in conjunction with other help-seeking promotion approaches to interrupt high-risk trajectories before they lead to chronic maladjustment and risk for suicide.

Innovation and Impact: While there has been substantial attention to the importance of promoting Veterans' use of mental health care, the investigators are not aware of any broad, measurement-based effort to enhance Veterans' willingness to seek help for multiple areas of unmet need. In addition, most intervention strategies are targeted to the needs of Veterans with chronic patterns of functional impairment and poor health rather than Veterans who experience initial readjustment challenges as they adapt to post-military life. The current project is innovative in its evaluation of a self-administered, population-based approach to raise Veterans' awareness of areas in which they may benefit from additional support and to connect them with relevant resources. Given that MBTA may be most beneficial to Veterans who experience initial readjustment challenges as they adapt to post-military life, this intervention will be evaluated among Veterans who have recently left military service.

Specific Aim: Aim 1 is to refine MBTA based on input from VA stakeholders (n=6) and qualitative interviews with Veterans (n=12). A key focus of this aim is to determine the optimal approach for presenting results and recommended resources. Aim 2 is to evaluate the feasibility, acceptability, and preliminary effectiveness of MBTA in promoting Veterans' support-seeking by testing this intervention in a sample of 60 Veterans.

Methodology: The proposed work will be guided by established methods for intervention development and implementation that emphasize user-centered design principles and iterative cycles of refinement and pilot testing to enhance MBTA's effectiveness and scalability. After refining MBTA based on feedback from VA stakeholders and Veterans (Aim 1), a national sample of Veterans will be randomized to MBTA or an assessment-only condition in a pilot randomized controlled trial (RCT) (Aim 2). The MBTA assessment will be comprised of validated measures of Veterans' status, functioning, and satisfaction across life domains, along with well-established mental health screeners. Veterans in the MBTA condition will receive a user-friendly web-based report that summarizes areas of unmet need, as well as tailored recommendations for relevant resources. Feasibility and acceptability will be evaluated based on participation and completion rates, as well as satisfaction and usability ratings. The investigators will also examine preliminary evidence for effectiveness by comparing pre-post changes in support-seeking outcomes for Veterans in intervention and control conditions. Only quantitative results from this pilot study are presented in clinicaltrials.gov.

Next Steps/Implementation: This pilot study will inform a subsequent proposal for a fully powered RCT to confirm the effectiveness of MBTA and to evaluate strategies to promote its dissemination and implementation.

ELIGIBILITY:
Inclusion Criteria:

* having separated from active duty military service within the prior three years, but not the past three months (for whom not enough time may have gone by to adequately assess readjustment challenge)
* having a postal address in the U.S
* having access to the internet

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawne S Vogt, PhD BA, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were recruited through invitations via mail between November 2022 and December 2022. 500 invitations were mailed (25 were undeliverable). Forty-six veterans accessed the study website URL and consented to participate.
Pre-assignment Details: Potential participants were randomly assigned to a group prior to mailing (250 to Intervention Group arm and 250 to Active Control Group arm)
Groups:
- Intervention Group: MBTA, MBTA satisfaction measures, and other assessment measures at T1; MBTA and other assessment measures at T2
  Measurement-Based Transition Assistance (MBTA) asks Veterans about their well-being and then provides Veterans with individualized feedback on areas in which they would benefit from additional support with regard to their health, vocational, financial, and social circumstances, along with personalized recommendations for relevant programs, services, and supports.
- Active Control Group: assessment measures only at T1; MBTA, MBTA satisfaction measures, and other assessment measures at T2
  Measurement-Based Transition Assistance (MBTA) asks Veterans about their well-being and then provides Veterans with individualized feedback on areas in which they would benefit from additional support with regard to their health, vocational, financial, and social circumstances, along with personalized recommendations for relevant programs, services, and supports.
Period: Overall Study
Arm/Group | Intervention Group | Active Control Group
Started | 27 | 19
Completed (completed both baseline and follow-up) | 15 | 10 (10 Veterans in the Active Control group completed MBTA at T2)
Not Completed | 12 | 9
Not completed — Lost to Follow-up | 9 | 9
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: Baseline participants are those that provided data in baseline. It does not include participants that consented to participate but then did not provide any data
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Active Control Group | Total
Number analyzed (Participants) | 24 | 19 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Not all participants provided data related to their age
  years
    number analyzed (Participants) | 17 | 19 | 36
    (all) | 41.71 (11.12) | 35.16 (8.73) | 38.25 (10.33)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Not all participants provided data related to their gender
  Participants
    Male: number analyzed (Participants) | 21 | 19 | 40
    Male | 15 | 13 | 28
    Female: number analyzed (Participants) | 21 | 19 | 40
    Female | 5 | 6 | 11
    Other or prefer not to say: number analyzed (Participants) | 21 | 19 | 40
    Other or prefer not to say | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 20 | 14 | 34
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 4 | 9
  White | 17 | 12 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 19 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Assessed for the Feasibility of Study Procedures
Description: Participation in the study will be evaluated to assess feasibility of the study procedures. To determine feasibility, at the end of data collection the investigators will calculate the following:
  1. Percentage of veterans who enroll in the study out of those invited (baseline; T1)
  2. Percentage of veterans who complete both T1 and T2 surveys (baseline [T1] and three-month follow-up [T2] data)
  3. Percentage of veterans who access the MBTA assessment (baseline [T1] for intervention group; three-month follow-up [T2] for active control group)
  4. Percentage of veterans who complete the MBTA assessment (baseline [T1] for intervention group; three-month follow-up [T2] for active control group)
  5. Percentage of veterans who review the personalized well-being report (baseline [T1] for intervention group; three-month follow-up [T2] for active control group)
Time Frame: baseline (T1) and three-month follow-up (T2)
Population: 500 letters mailed; number analyzed varies per row because of number of eligible participants within each category/row
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Group: MBTA, MBTA satisfaction measures, and other assessment measures at T1 (baseline); MBTA and other assessment measures at T2 (three-month follow-up)
  Measurement-Based Transition Assistance (MBTA) asks Veterans about their well-being and then provides Veterans with individualized feedback on areas in which they would benefit from additional support with regard to their health, vocational, financial, and social circumstances, along with personalized recommendations for relevant programs, services, and supports.
Arm/Group | Intervention Group | Active Control Group
Number analyzed (Participants) | 250 | 250
Participants
  Percent of veterans who enroll in the study out of those invited (T1; baseline) | 27 | 19
  Percent of veterans who complete both baseline and three-month follow-up surveys (T1 and T2 data): number analyzed (Participants) | 24 | 19
  Percent of veterans who complete both baseline and three-month follow-up surveys (T1 and T2 data) | 15 | 10
  Percent who access MBTA assessment (Intervention: baseline; Active Control: three-month follow-up): number analyzed (Participants) | 24 | 10
  Percent who access MBTA assessment (Intervention: baseline; Active Control: three-month follow-up) | 22 | 10
  Percent who complete MBTA assessment (Intervention: baseline; Active Control: three-month follow-up): number analyzed (Participants) | 22 | 10
  Percent who complete MBTA assessment (Intervention: baseline; Active Control: three-month follow-up) | 21 | 10
  Percent who review the personal report (Intervention:baseline; Active Control:three-month follow-up): number analyzed (Participants) | 21 | 10
  Percent who review the personal report (Intervention:baseline; Active Control:three-month follow-up) | 21 | 10

2. Primary Outcome: Satisfaction With MBTA Tool
Description: For the intervention group at the baseline assessment (T1), the investigators assessed satisfaction with the MBTA tool with items developed specifically for this pilot study. T1 (baseline) was the only timeframe these questions were administered for this group). The investigators asked open-ended questions such as: What did you like about the tool? What did you not like about the tool? Is there anything you would change about the tool?
Time Frame: baseline assessment (T1 only for intervention group)
Population: 16 Veterans in the intervention group provided data for open-ended questions at T1 (baseline). T1 (baseline) was the only timeframe when these questions were administered for this group.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 16
Participants
  Provided positive feedback about MBTA prototype | 14
  Provided a critique about MBTA prototype | 5
  Provided constructive feedback about MBTA prototype | 4

3. Primary Outcome: Satisfaction With MBTA Tool
Description: For the active control group, they were asked at the three-month follow-up (T2) their satisfaction with the MBTA tool with items developed specifically for this pilot study. T2 (three-month follow-up) was the only timeframe these questions were administered for this group). The investigators asked open-ended questions such as: What did you like about the tool? What did you not like about the tool? Is there anything you would change about the tool?
Time Frame: three-month follow-up (T2 only for active control group)
Population: 7 Veterans in the active control group provided data for open-ended questions at T2 (three-month follow-up). T2 (three-month follow-up) was the only timeframe when these questions were administered for this group
Measure: Count of Participants; unit: Participants
Groups:
- Active Control Group: assessment measures only at T1 (baseline); MBTA, MBTA satisfaction measures, and other assessment measures at T2 (three-month follow-up)
  Measurement-Based Transition Assistance (MBTA) asks Veterans about their well-being and then provides Veterans with individualized feedback on areas in which they would benefit from additional support with regard to their health, vocational, financial, and social circumstances, along with personalized recommendations for relevant programs, services, and supports.
Arm/Group | Active Control Group
Number analyzed (Participants) | 7
Participants
  Provided positive feedback about MBTA prototype | 7
  Provided a critique about MBTA prototype | 3
  Provided constructive feedback about MBTA prototype | 2

4. Secondary Outcome: University of Rhode Island Change Assessment Scale (URICA) - Readiness to Change
Description: The investigators administered the University of Rhode Island Change Assessment Scale (URICA; DiClemente et al., 2004) to measure movement in the stages of change. Questions in the URICA were slightly modified to focus on well-being. To score the URICA, the investigators will calculate a readiness to change score based on the four stages of change (precontemplation, contemplation, action, and maintenance). The investigators will calculate means for precontemplation responses, contemplation responses, action responses and maintenance responses and subtract the mean from the precontemplation score from the summation of the other three stages. This sum score represents an individual's readiness to change. Possible readiness to change scores range from -2 to +14, with higher scores indicating higher levels of readiness to change.
Time Frame: measured at T1(baseline) and T2 (three-month follow-up) for the intervention group and active control group; estimates reported below are three-month follow-up adjusted mean scores
Population: An overall readiness to change score was calculated at T1 (baseline) and T2 (three-month follow-up). Using ANCOVAs, data values represent three-month follow-up adjusted mean scores after controlling for baseline scores and age.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Group | Active Control Group
Number analyzed (Participants) | 8 | 9
score on a scale | 11.20 (0.72) | 10.69 (0.68)
Statistical Analysis 1: Comparison: Intervention Group vs Active Control Group; Test type: Superiority; p = .617, ANCOVA; Partial Eta Squared (effect size) = .020

5. Secondary Outcome: Stages Algorithm
Description: The investigators administered the Stages Algorithm (DiClemente et al., 1991) to measure movement in the stages of change from baseline to the three-month follow-up. Questions were modified slightly to assess for willingness to work on resolving problems or challenges related to areas of well-being (i.e., mental health/emotional well-being, physical health, vocation, social life, and finances). This measure is designed as a decision tree based on reported challenges, and is scored based on where participants fall within the decision tree. It classifies participants according to the following stages of change: precontemplation, contemplation, preparation, action, and maintenance stages.
Time Frame: measured at T1 (baseline) and T2 (three-month follow-up) for the intervention group and active control group; challenges reported are from baseline (T1) and if they were were taking action to address these challenges are data from three-month follow-up
Population: Data were collected for intervention and active control group at baseline and three-month follow-up. Among participants who identified a challenge within a domain. Then within that subgroup of those with challenges, we examined the number that moved forward at least one stage/were taking action to work on their challenges between baseline (T1) and the three-month follow-up (T2).
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Group: MBTA, MBTA satisfaction measures, and other assessment measures at T1 (baseline); MBTA and other assessment measures at T2 (three-month follow-up)
- Active Control Group: assessment measures only at T1 (baseline); MBTA, MBTA satisfaction measures, and other assessment measures at T2 (three-month follow-up)
Arm/Group | Intervention Group | Active Control Group
Number analyzed (Participants) | 15 | 10
Participants
  Vocation (reported challenges at T1; baseline) | 7 | 5
  Vocation(of those reporting challenges at T1, # that were taking action to work on challenges at T2): number analyzed (Participants) | 7 | 5
  Vocation(of those reporting challenges at T1, # that were taking action to work on challenges at T2) | 7 | 5
  Finances (reported challenges at T1; baseline) | 5 | 3
  Finances(of those reporting challenges at T1, # that were taking action to work on challenges at T2): number analyzed (Participants) | 5 | 3
  Finances(of those reporting challenges at T1, # that were taking action to work on challenges at T2) | 5 | 2
  Social (reported challenges at T1; baseline) | 11 | 5
  Social (of those reporting challenges at T1, # that were taking action to work on challenges at T2): number analyzed (Participants) | 11 | 5
  Social (of those reporting challenges at T1, # that were taking action to work on challenges at T2) | 10 | 4
  Mental Health (reported challenges at T1; baseline) | 9 | 7
  Mental Health(of those with challenges at T1, # that were taking action to work on challenges at T2): number analyzed (Participants) | 9 | 7
  Mental Health(of those with challenges at T1, # that were taking action to work on challenges at T2) | 7 | 6
  Physical Health (reported challenges at T1; baseline) | 13 | 7
  Physical Health(of those with T1 challenges, # that were taking action to work on challenges at T2): number analyzed (Participants) | 13 | 7
  Physical Health(of those with T1 challenges, # that were taking action to work on challenges at T2) | 10 | 7

6. Secondary Outcome: Theory of Planned Behavior Constructs
Description: The investigators used Theory of Planned Behavior Questionnaire (Ajzen, 1991) to assess movement from baseline to the three-month follow-up in the constructs from the theory of planned behavior (intention, attitude toward the behavior, subjective norm, perceived behavioral control). Questions were slightly modified to focus on well-being. The investigators scored each of the aforementioned constructs/subscales separately. For each subscale, the investigators calculated the the mean of the items. Scores could range from 1 to 7 with higher scores indicating a more positive response.
Time Frame: measured at T1 (baseline) and T2 (three-month follow-up) for the intervention group and active control group; estimates reported below are three-month follow-up adjusted mean scores
Population: Scores were calculated at T1 (baseline) and T2 (three-month follow-up) for intervention and active control group. Scores could range from 1 to 7 with higher scores indicating a more positive response. Number of participants analyzed for each row varies based on the number of participants that provided data for that construct at both time points. Using ANCOVAs, data values represent three-month follow-up adjusted mean (follow-up) scores after controlling for baseline scores and age.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Group | Active Control Group
Number analyzed (Participants) | 11 | 10
score on a scale
  Intentions | 4.95 (0.35) | 5.61 (0.36)
  Attitudes: number analyzed (Participants) | 10 | 10
  Attitudes | 5.97 (0.31) | 6.03 (0.31)
  Social norms: number analyzed (Participants) | 11 | 9
  Social norms | 5.14 (0.33) | 4.68 (0.36)
  Perceived behavioral control | 5.53 (0.32) | 5.05 (0.34)
Statistical Analysis 1: Comparison: Intervention Group vs Active Control Group; Null hypothesis: Intervention and active control group intention follow-up means are equal when controlling for covariates (i.e., baseline intention scores and age); Test type: Superiority; p = .214, ANCOVA; Partial Eta Squared (effect size) = .089
Statistical Analysis 2: Comparison: Intervention Group vs Active Control Group; Null hypothesis: Intervention and active control group attitude follow-up means are equal when controlling for covariates (i.e., baseline attitude scores and age); Test type: Superiority; p = .894, ANCOVA; Partial Eta Squared (effect size) = .001
Statistical Analysis 3: Comparison: Intervention Group vs Active Control Group; Null hypothesis: Intervention and active control group social norms follow-up means are equal when controlling for covariates (i.e., baseline social norms scores and age); Test type: Superiority; p = .359, ANCOVA; Partial Eta Squared (Effect Size) = .053
Statistical Analysis 4: Comparison: Intervention Group vs Active Control Group; Null hypothesis: Intervention and active control group perceived behavioral control follow-up means are equal when controlling for covariates (i.e., baseline perceived behavioral control scores and age); Test type: Superiority; p = .322, ANCOVA; Partial Eta Squared (Effect Size) = .058

7. Secondary Outcome: Attitudes Toward Seeking Professional Psychological Help-Short Form
Description: The investigators assessed movement in support seeking perceptions from baseline (T1) to the three-month follow-up (T2) with the Attitudes Toward Seeking Professional Psychological Help - Short Form scale (Picco et al., 2016). Questions were slightly modified to focus on seeking support to address well-being challenges and problems. To calculate a total score, items 2, 4, 8, 9, and 10 were reverse scored. Scores were then summed together, with higher scores indicating more positive attitudes toward seeking professional help. Scores could range range for 0-30.
Time Frame: as for outcome 6
Population: Possible scores ranged from 0 to 30, with higher scores indicating more positive attitudes toward seeking professional help. Using ANCOVAs, data values represent three-month follow-up adjusted mean (follow-up) scores after controlling for baseline scores and age
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention Group | Active Control Group
Number analyzed (Participants) | 11 | 10
score on a scale | 19.24 (0.95) | 19.04 (1.00)
Statistical Analysis 1: Comparison: Intervention Group vs Active Control Group; Test type: Superiority; p = .891, ANCOVA; Partial Eta Squared (effect size) = .001

8. Secondary Outcome: Support-Seeking Actions to Improve Well-Being
Description: For the intervention group, the investigators assessed support seeking behavior with items developed specifically for this pilot study at T2 (three-month follow-up). Questions asked about the extent to which the tool has helped increase awareness about well-being related challenges or problems, the extent to which the tool has helped encourage improving well-being related problems or challenges, and which types of resources the participant has used since using the tool. Items were examined separately. A response of moderately or higher on the two Likert scale items was considered a positive response.
Time Frame: Measured at T2 (three-month follow-up) for intervention group only
Population: 15 veterans in the intervention group provided data for support-seeking actions at T2 (three-month follow-up); number of participants analyzed is different because type of service percentage applies only to those that used services (n=10). These measures were only administered to the intervention group at T2 (three-month follow-up). These measures were not administered to the active control group at either time point.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Group: MBTA, MBTA satisfaction measures, and other assessment measures at T1; MBTA and other assessment measures at T2
Arm/Group | Intervention Group
Number analyzed (Participants) | 15
Participants
  Reported MBTA prototype increased awareness about their well-being related challenges or problems | 6
  Reported MBTA prototype helped encourage them to improve well-being related problems or challenges | 7
  Reported using a resource/service (not previously using before study) as a result the MBTA prototype | 10
  Used a mental health resource/service: number analyzed (Participants) | 10
  Used a mental health resource/service | 5
  Used a financial resource/service: number analyzed (Participants) | 10
  Used a financial resource/service | 2
  Used a health behavior resource/service: number analyzed (Participants) | 10
  Used a health behavior resource/service | 1
  Used other general health resource/service: number analyzed (Participants) | 10
  Used other general health resource/service | 1
  Used a resource/service related to their social life: number analyzed (Participants) | 10
  Used a resource/service related to their social life | 1
  Used a resource/service under an 'other' category: number analyzed (Participants) | 10
  Used a resource/service under an 'other' category | 3
  Used a vocation-related resource/service: number analyzed (Participants) | 10
  Used a vocation-related resource/service | 0

ADVERSE EVENTS:
Time Frame: 3 months (from baseline to 3-month follow-up)
Description: The 34 participants listed in the MBTA Intervention group represent all participants that received the MBTA intervention at any time point during the study (24 participants in the intervention group accessed MBTA at baseline + 10 participants from the Active Control group accessed MBTA at the three-month follow-up). The 9 participants listed in the Active Control Group did not access MBTA because they only participated in the study at baseline which they were unable to access MBTA at that time.
Groups:
- Intervention Group: MBTA, MBTA satisfaction measures, and other assessment measures at T1 (baseline); MBTA and other assessment measures at T2 (three-month follow-up)
  Measurement-Based Transition Assistance: Measurement-Based Transition Assistance (MBTA) provides Veterans with individualized feedback on areas in which they would benefit from additional support with regard to their health, vocational, financial, and social circumstances, along with personalized recommendations for relevant programs, services, and supports.
Arm/Group | Intervention Group | Active Control Group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/9
Other Adverse Events (participants affected / at risk) | 0/34 | 0/9

LIMITATIONS AND CAVEATS:
The number of veterans that enrolled in this pilot study was lower than expected which resulted in the study being underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT05384171/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT05384171/ICF_001.pdf